CLINICAL TRIAL: NCT00584428
Title: High Dose Chemotherapy With Autologous Bone Marrow Transplantation in the Treatment of Metastatic Breast Cancer
Brief Title: High Dose Chemo With Autologous BMT for Treatment of Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Stephenson Cancer Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU 9206; OU 9206
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Cancer Treatment; Breast Cancer Treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: High-Dose Chemo with Autologous BMT

INTERVENTIONS:
Procedure: High-Dose Chemo with Autologous BMT — Carboplatin/VP-16/Cytoxan for women 18-59 and Carboplatin/Thiotepa/Cytoxan for women 60-70

SUMMARY:
To evaluate the response rate and the response duration of high dose chemotherapy with autologous bone marrow transplantation as intensification following induction chemotherapy in metastatic breast cancer and to evaluate prospectively the subdivision of patients with metastatic breast cancer according to prognostic groups.

DETAILED DESCRIPTION:
There are 2 phases to this study: 1) Induction- which consists of the administration of chemotherapeutic drugs- at the end of this phase if the cancer has responded, bone marrow will be collected and frozen untol ready for re-infusion; 2) 2nd phase- involves high-doses of chemotherapy followed by infusion of bone marrow cells

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of breast cancer
* Age 18-70
* Breast cancer at first clinical evidence of metastatic disease
* Must have objectively measurable or evaluable disease or be in complete remission

Exclusion Criteria:

* Previous diagnosis of another invasive carcinaom within 10 years (except skin cancer)
* CNS involvement

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 1992-06; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Once 10 patients enrolled in the study ar followed for at least 6 months, a preliminary analysis of the data will occur. | Undetermined

SECONDARY OUTCOMES:
No secondary outcomes | Undetermined

CONTACTS AND LOCATIONS:
Overall Officials: George Selby, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States